CLINICAL TRIAL: NCT07387744
Title: Assessing Ambulatory and Non-ambulatory Community Mobility in People With Lower Limb Amputation.
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Virginia Commonwealth University (Other)
Collaborators: National Center for Advancing Translational Sciences (NCATS) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: HM20033204; K12TR004364 (NIH)
Record Dates: First submitted 2026-01-27; First posted 2026-02-04 (Actual); Last update posted 2026-02-04 (Actual); Status verified 2026-01

CONDITIONS: Amputation
Keywords: Lower Limb Amputation (LLA); Global Positioning System (GPS)

STUDY DESIGN:
Intervention Model Description: Prospective cohort study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Lower Limb Amputation (LLA) Participants (Experimental): People with lower limb amputation will be targeted as this is the population of interest for this study.
  Interventions: Other: Clinical Descriptive Measures related to amputation collected; Other: GPS device education/distributed; Other: activPAL device education/distributed; Other: Questionnaire Assessments completed

INTERVENTIONS:
Other: Clinical Descriptive Measures related to amputation collected — On Visit 1 (baseline) Clinical measures will be collected including: Amputation level, date of amputation, amputation etiology, assistive device used and Medicare K level. The measures are intended for demographic and descriptive use.
Other: GPS device education/distributed — The QStarz GPS data logger will be worn for all waking hours (from 8 am to 8 pm or beyond if awake), even on days they do not plan to leave home. The device is worn on a belt, in a pocket, or in a bag/pouch. Education on how to wear, maintain and charge the device will be provided.
Other: activPAL device education/distributed — Participants will wear a thigh-mounted activPAL micro accelerometer on their non-amputated limb (or longest residual limb if bilateral amputation). The activPAL sensor is small and lightweight, secured to the thigh with a waterproof dressing, and participants are instructed to wear it at all times (including sleep) unless swimming. Education on how to wear the device will be provided.
Other: Questionnaire Assessments completed — For visit #1 only, the following assessments will be completed: World Health Organization Quality of Life Brief Assessment (WHOQOL-BREF), Prosthesis Evaluation Questionnaire - Mobility subscale, Locomotor Capabilities Index, Modified telephone interview for cognitive status, Life Space Assessment, Houghton Scale, World health organization disability assessment schedule 2.0 (WHODAS) and Activities-specific balance confidence scale

SUMMARY:
Mobility is a fundamental aspect of daily life, enabling individuals to participate in social, occupational, and recreational activities. Community mobility, defined as movement in environments outside the home, is particularly important for quality-of-life. Following lower limb amputation (LLA), mobility limitations are common and persistent. With rehabilitation and prosthetic training, many regain the ability to ambulate but results vary as only 25 - 58% of patients regain ambulatory ability and less than half of those who become ambulatory achieve sufficient ability to walk in community settings. As a result, ~40% of people with LLA are ambulatory but also use wheeled mobility (e.g., wheelchair, scooter) for some or all of their community mobility tasks. To date, the complementary role of wheeled and ambulatory mobility in maximizing community mobility has been overlooked, with clinical research overwhelmingly focused on assessing and improving ambulatory ability despite its impracticality for many community settings.

DETAILED DESCRIPTION:
Poor understanding of the multiple mobility modes used by people with lower limb amputation (LLA) is a likely contributor high rates of self-reported disability, poor social engagement, and lower quality of life. Understanding mobility patterns in this population is essential for developing targeted interventions, optimizing assistive technologies, and improving overall community mobility. This study addresses three limitations in rigor of prior research on community mobility in people with LLA: 1) minimal use of objectively-monitored community mobility, 2) unknown contexts of ambulatory and wheeled mobility behaviors, 3) unclear relationship between patient and clinical factors influencing mode of community mobility.

ELIGIBILITY:
Inclusion Criteria:

* Unilateral or bilateral major lower limb amputation (e.g., proximal to or through the ankle joint)
* >6 months since LLA Fitted with a prosthetic limb
* Fitted with a prosthetic limb
* Use a wheelchair or scooter for mobility for part of a day at least once per week

Exclusion Criteria:

* Unstable heart condition (including unstable angina, uncontrolled cardiac dysrhythmia, acute myocarditis, hypertension, and acute pericarditis)
* Acute systemic infection Prisoner or institutionalized such that self-determined mobility is restricted
* Prisoner or institutionalized such that self-determined mobility is restricted
* Decisionally challenged individuals (Modified Telephone Interview for Cognitive Status score ≤24)
* Undergoing active cancer treatment
* Participating in prosthetic rehabilitation
* Clinical discretion of the principal investigator to exclude patients who are determined to be unsafe and/or inappropriate to participate in the protocol
* Inability to communicate verbally in English

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2026-03 (Estimated); Primary Completion 2027-08 (Estimated); Study Completion 2027-08 (Estimated)

PRIMARY OUTCOMES:
World Health Organization Quality of Life Brief Assessment (WHOQOL-BREF) | Visit 1 (Baseline) only/no repeated measures
  The (WHOQOL-BREF) is a standardized assessment of an individual's perceived quality of life across physical, psychological, social, and environmental domains. The WHOQOL-BREF is a widely used, 26-item self-report questionnaire from the World Health Organization that assesses an individual's Quality of Life (QOL) across four core domains: Physical Health, Psychological Health, Social Relationships, and Environment, plus two additional items for overall QOL and health. It's a brief, cross-culturally valid tool, derived from the longer WHOQOL-100, providing reliable data for research and clinical use by asking about experiences over the past two weeks on a 5-point scale. Higher scores (closer to 100) indicate better quality of life within that domain. Not evaluating any change, just a snapshot in time at Visit 1.
Prosthesis Evaluation Questionnaire - Mobility subscale | Visit 1 (Baseline) only/no repeated measures
  The Prosthesis Evaluation Questionnaire - Mobility subscale, captures a person's self reported ability to move and perform daily activities while using their prosthesis. It uses a 5-point ordinal scale (0-4). 0: Not able or hardly able to 4: No problem or almost fully able. The total scale ranges from 0 to 48. A higher score indicates more mobility. Not evaluating any change, just a snapshot in time at Visit 1.
Locomotor Capabilities Index | Visit 1 (Baseline) only/no repeated measures
  The Locomotor Capabilities Index measures a person's perceived ability to perform everyday mobility tasks using their prosthesis. The Locomotor Capabilities Index (LCI) is a validated, 14-item self-administered questionnaire used to assess the walking ability and independence of lower-limb amputees using a prosthesis. It evaluates a patient's perceived capability-what they believe they can do-rather than their actual everyday performance. The max score is 42. Not evaluating any change, just a snapshot in time at Visit 1.
Modified telephone interview for cognitive status | Visit 1 (Baseline) only/no repeated measures
  The Modified telephone interview for cognitive status is a brief, 13-item structured screening of global cognitive function suitable for remote administration. It is widely used in large-scale epidemiological studies and clinical practice to differentiate between normal aging, mild cognitive impairment (MCI), and dementia. Scores on the TICS-M range from 0 to 50, with higher scores indicating better cognitive health. Not evaluating any change, just a snapshot in time at Visit 1.
Life Space Assessment | Visit 1 (Baseline) only/no repeated measures
  The Life Space Assessment quantifies how far, how often, and how independently a person moves through their environment in daily life. A score of 60 or below is the standard threshold indicating restricted life-space.
  Assessment calculation:
  Frequency: How often did they reach this level (1 = <1x/week, 2 = 1-3x/week, 3 = 4-6x/week, 4 = daily)? Independence: Did they require help (1 = personal assistance, 1.5 = equipment only, 2
  = no equipment or personal assistance)? The Composite LSA Score (0-120) is calculated by multiplying the Level (1-5) × Frequency (1-4) × Independence (1-2) for each of the five levels and summing the results.
  Not evaluating any change, just a snapshot in time at Visit 1.
Houghton Scale | Visit 1 (Baseline) only/no repeated measures
  The Houghton Scale assesses a person's confidence and ability in using their prosthesis safely and effectively during everyday mobility tasks. The Houghton Scale is a self-administered, 4-item questionnaire used to assess the functional use of a prosthesis by individuals with lower-limb amputations.It measures how often a patient wears their prosthesis, the types of activities they perform with it, and their perceived stability in various outdoor environments. Total scores range from 0 to 12, with higher scores indicating greater prosthesis use and independence. Not evaluating any change, just a snapshot in time at Visit 1.
World health organization disability assessment schedule 2.0 (WHODAS) | Visit 1 (Baseline) only/no repeated measures
  The World health organization disability assessment schedule 2.0 (WHODAS) evaluates how health conditions impact a person's functioning and participation across major life domains over the past 30 days. Items are rated on a 5-point Likert scale: None (0), Mild (1), Moderate (2), Severe (3), and Extreme or Cannot Do (4). While no universal "cut-off" exists, scores placing a patient in the top 10% of the population distribution-roughly >10 for the 12-item simple score or >41 for the 36-item version-likely indicate significant impairment. Not evaluating any change, just a snapshot in time at Visit 1.
Activities-specific balance confidence scale | Visit 1 (Baseline) only/no repeated measures
  The Activities-specific balance confidence scale is a self-report instrument used to measure an individual's confidence in maintaining balance while performing 16 various daily activities. Unlike performance-based tests, it captures the patient's perceived ability to avoid falling or becoming unsteady.Patients rate their confidence for each item on a scale from 0% (no confidence) to 100% (complete confidence). The higher the score,the higher the function and physical activity (range > 80% high function, 50% - 80% moderate function and < 50% low function. Not evaluating any change, just a snapshot in time at Visit 1.
GPS Outcomes (spatial and temporal metrics of community mobility):Total Distance Traveled (m) | Data collected visit #1 through visit #2, data collected for 10-21 days, downloaded on Visit #2
  On visit #1 subjects are provided with the device and education. The device will be worn 10-21 days (based on scheduling logistics). Total Distance Traveled data will be downloaded and reported in meters (m) as an aggregate mean.
GPS Outcomes (spatial and temporal metrics of community mobility): Average movement speed (km/hr) | Data collected visit #1 through visit #2, data collected for 10-21 days, downloaded on Visit #2
  On visit #1 subjects are provided with the device and education. The device will be worn 10-21 days (based on scheduling logistics). Average Movement data will be downloaded and reported in (km/hr) as an aggregate mean
GPS Outcomes (spatial and temporal metrics of community mobility): Size of movement area (km2) | Data collected visit #1 through visit #2, data collected for 10-21 days, downloaded on Visit #2
  On visit #1 subjects are provided with the device and education. The device will be worn 10-21 days (based on scheduling logistics). Size of movement area data will be downloaded and reported in (km2) as an aggregate mean
GPS Outcomes (spatial and temporal metrics of community mobility): Percentage of time spent outside the home | Data collected visit #1 through visit #2, data collected for 10-21 days, downloaded on Visit #2
  On visit #1 subjects are provided with the device and education. The device will be worn 10-21 days (based on scheduling logistics). Percentage of time spent outside the home data will be downloaded and reported in minutes as an aggregate mean.
GPS Outcomes (spatial and temporal metrics of community mobility): Mean and median distance from home | Data collected visit #1 through visit #2, data collected for 10-21 days, downloaded on Visit #2
  On visit #1 subjects are provided with the device and education. The device will be worn 10-21 days (based on scheduling logistics). Mean and median distance from home will be downloaded and reported in (m) as an aggregate mean.
GPS Outcomes (spatial and temporal metrics of community mobility): Number of locations visited | Data collected visit #1 through visit #2, data collected for 10-21 days, downloaded on Visit #2
  On visit #1 subjects are provided with the device and education. The device will be worn 10-21 days (based on scheduling logistics). The number of locations visited will be downloaded and reported as a total number
GPS Outcomes (spatial and temporal metrics of community mobility): Max distance from home (km) | Data collected visit #1 through visit #2, data collected for 10-21 days, downloaded on Visit #2
  On visit #1 subjects are provided with the device and education. The device will be worn 10-21 days (based on scheduling logistics). Max distance from home (km) will be downloaded and reported as an aggregate mean.
GPS Outcomes (spatial and temporal metrics of community mobility): Frequency of out-of-home trips | Data collected visit #1 through visit #2, data collected for 10-21 days, downloaded on Visit #2
  On visit #1 subjects are provided with the device and education. The device will be worn 10-21 days (based on scheduling logistics). Frequency of out-of-home trips data will be downloaded and reported as an overall total number.
GPS Outcomes (spatial and temporal metrics of community mobility): Time and distance on foot | Data collected visit #1 through visit #2, data collected for 10-21 days, downloaded on Visit #2
  On visit #1 subjects are provided with the device and education. The device will be worn 10-21 days (based on scheduling logistics). Time and distance on foot will be downloaded and reported as an aggregate mean
activPAL Accelerometry: Daily duration (in minutes) of sitting, standing, and stepping | Data collected visit #1 through visit #2, data collected for 10-21 days, downloaded on Visit #2
  On visit #1 subjects are provided with the device and education. The device will be worn 10-21 days (based on scheduling logistics). Daily duration (in minutes) of sitting, standing, and stepping will be downloaded and reported as an aggregate mean.
activPAL Accelerometry: Daily step count | Data collected visit #1 through visit #2, data collected for 10-21 days, downloaded on Visit #2
  On visit #1 subjects are provided with the device and education. The device will be worn 10-21 days (based on scheduling logistics). Daily step count data will be downloaded and reported as an aggregate mean.
activPAL Accelerometry: Daily walking bouts stepping cadence | Data collected visit #1 through visit #2, data collected for 10-21 days, downloaded on Visit #2
  On visit #1 subjects are provided with the device and education. The device will be worn 10-21 days (based on scheduling logistics). The stepping cadence of daily walking bouts will be downloaded and reported as an aggregate mean.

CONTACTS AND LOCATIONS:
Overall Officials: Paul Kline, Principal Investigator — Virginia Commonwealth University
Locations (1):
- Virginia Commonwealth University, Richmond, Virginia, United States